CLINICAL TRIAL: NCT05611372
Title: Efficacy and Safety of Rasagiline in Prodromal Parkinson's Disease
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No suitable recruitment
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Beijing Tiantan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Jiangsu Province Nanjing Brain Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Huashan Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Guizhou Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); West China Hospital (Other); Sir Run Run Shaw Hospital (Other); The Affiliated Hospital of Hangzhou Normal University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Qilu Hospital of Shandong University (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAHZJU_RBD
Record Dates: First submitted 2022-11-06; First posted 2022-11-10 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2022-11

CONDITIONS: REM Sleep Behavior Disorder; Parkinson Disease; Synucleinopathies
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease; Synucleinopathies | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Intervention (Experimental): 0-52 week: rasagiline 1 mg/day
  Interventions: Drug: Rasagiline
- Delayed Intervention (Active Comparator): 0-26 week: palcebo 1mg/day 27-52 week: rasagiline 1mg/day
  Interventions: Drug: Rasagiline

INTERVENTIONS:
Drug: Rasagiline — 1 mg rasagiline

SUMMARY:
To investigate whether a year of rasagiline may reduce the progression from idiopathic REM sleep behavior disorder (RBD) to Parkinson's disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* PSG confirmed RBD with subtle motor symptoms (4≤MDS-UPDRS-III≤10 at baseline)
* no clinical diagnosis of Parkinson's disease or dementia at baseline
* age 30-75
* no concomitant or previous use of any other anti-parkinson medications
* provide written informed consent

Exclusion Criteria:

* diagnosed with secondary parkinsonism (eg., drug-induced, vascular, psychogenic)
* secondary RBD (eg., drug-induced, immune-mediated)
* nervous system comorbidities (eg., stroke, epilepsy, encephalitis)
* severe psychiatric comorbidities
* allergic to rasagiline
* severe systemic diseases (eg., end-stage kidney disease, liver failure)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival time | 3 years after starting rasagiline treatment
  Not diagnosed as any of the synucleinopathies (Parkinson's disease; dementia with lewy body; multiple system atrophy)

SECONDARY OUTCOMES:
Striatal dopaminergic innervation | 0-3 years after starting rasagiline treatment
  Striatal binding ratio from DAT-Scan
MDS-UPDRS-III | 0-3 years after starting rasagiline treatment
MoCA | 0-3 years after starting rasagiline treatment
MMSE | 0-3 years after starting rasagiline treatment
HAMA | 0-3 years after starting rasagiline treatment
HAMD | 0-3 years after starting rasagiline treatment
RBDQ-HK | 0-3 years after starting rasagiline treatment
PSQI | 0-3 years after starting rasagiline treatment
PDQ39 | 0-3 years after starting rasagiline treatment
SCOPA-AUT | 0-3 years after starting rasagiline treatment

CONTACTS AND LOCATIONS:
Overall Officials: Baorong Zhang, MD, Principal Investigator — Second Affiliated Hospital, Zhejiang University, China

IPD SHARING:
Plan to Share IPD: No